CLINICAL TRIAL: NCT05830656
Title: Recovering From Work Through Nature Experiences - Heading to the Forest or a Virtual Forest?
Brief Title: Hybrid- Nature: Recovering From Work Through Nature Experiences
Acronym: HybridNature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JAMK University Of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: JAMKUAS_Hybridnature
Record Dates: First submitted 2023-01-26; First posted 2023-04-26 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Physiological Recovery; Psychological Recovery; Restorative Experiences
Keywords: Recovery; Nature; Employees; Work stress; Occupational well-being; Virtual Reality
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control, Then exposure to nearby nature, Then exposure to virtual nature (Experimental): During the first week, the participants continue their normal routine at work and in leisure time. On the second week, the participants visit a nearby natural area after finishing their workday on three days (Tuesday, Wednesday, and Thursday). On the third week, the participants watch virtual nature videos with Virtual Reality (VR) goggles after finishing their workday on three days (Tuesday, Wednesday, and Thursday).
  Interventions: Behavioral: Exposure to nearby nature; Behavioral: Exposure to virtual nature
- Control, Then exposure to virtual nature, Then exposure to nearby nature (Experimental): During the first week, the participants continue their normal routine at work and in leisure time. On the second week, the participants watch virtual nature videos with Virtual Reality (VR) goggles after finishing their workday on three days (Tuesday, Wednesday, and Thursday). On the third week, the participants visit a nearby natural area after finishing their workday on three days (Tuesday, Wednesday, and Thursday).
  Interventions: Behavioral: Exposure to nearby nature; Behavioral: Exposure to virtual nature

INTERVENTIONS:
Behavioral: Exposure to nearby nature — Participants spend a minimum of 20 minutes in their favourite place in nearby nature.
Behavioral: Exposure to virtual nature — Participants spend a minimum of 20 minutes watching virtual nature videos.

SUMMARY:
The research examines employees' recovery from work stress during visits in nearby nature and when viewing virtual nature with Virtual Reality (VR) goggles. The research provides information on the physiological and psychological recovery of employees who do remote or hybrid work. Recovery is analysed with qualitative and quantitative methods including Firstbeat Life measurements, surveys and interviews. The results can be used in workplaces to develop operating models to promote well-being in remote and hybrid work. The research generates new understanding on how employees' recovery can be supported by means of virtual nature tourism services.

DETAILED DESCRIPTION:
An intervention study with a cross-over research design will be conducted among a sample of 60 employees who do remote or hybrid work. The intervention phase lasts in total of four weeks. During the first week (control phase), the participants continue their daily routine as normal. During the second week of the intervention, a half of the participants are randomised to visit a nearby natural area after finishing work (exposure to nearby nature). The other half of the participants are randomised to view virtual nature videos with VR goggles after finishing work (exposure to virtual nature). On the third week of the intervention, the participants complete nature exposure the other way around. That is, those participants who took part first in exposure to nearby nature will view virtual nature, and vice versa. On the fourth week of the intervention, the participants take part in a semi-structured focus group interview.

Recovering from work in nearby nature and virtual nature is examined through multidisciplinary perspectives of health, well-being, and tourism. The aim of the research is to find new ways of promoting work stress recovery, psychological detachment and restoration among employees when they are making the transition between work time and personal time. These research findings are particularly relevant for fields in which there has been a growing trend for remote or hybrid work. This research is funded by the Finnish Work Environment Fund (Project Number: 220076).

ELIGIBILITY:
Inclusion Criteria:

* Employees who do remote or hybrid work
* Able to communicate adequately in Finnish in order to participate

Exclusion Criteria:

* No exclusion criteria for study participation.
* Firstbeat Life analyses are only available for participants who identify themselves on the basis of biological sex of female or male.
* Firstbeat Life analyses might be unreliable for participants with some health-related issues (e.g., pacemaker, heart transplantation, complex cardiac disease, persistent atrial fibrillation or flutter, or uncontrolled thyroid disease) and therefore measurements will not be performed for them as a part of this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-16 (Actual)

PRIMARY OUTCOMES:
Psychological recovery | Three weeks
  Recovery Experience Questionnaire (REQ), the scores range from 1 to 5, a higher score refers to better psychological recovery.

SECONDARY OUTCOMES:
Restorative experiences | Three weeks
  Restorative Outcome Scale (ROS), the scores range from 1 to 7, a higher score refers to better restoration.
Work engagement | Three weeks
  Utrecht Work Engagement Scale (UWES), the scores range from 1 to 7, a higher score refers to higher work engagement.
Burnout | Three weeks
  Burnout Assessment Tool (BAT), the scores range from 1 to 5, a higher score refers to higher burnout.
Stress recovery | Three weeks
  A physiological measure of stress recovery balance, the scores range from 0 to 100, a higher score refers to better physiological stress recovery.
Sleep quality | Three weeks
  A physiological measure of the restorative effect of sleep, the scores range from 0 to 100, a higher score refers to better recovery during sleep.
Relax-Stress Intensity | Three weeks
  A physiological measure of the Relax-Stress Intensity (RSI), the scores range from -100 to 100, a higher score (+/- 100) refers to a stronger reaction.
Body resources | Three weeks
  A physiological measure of body resources, the scores range from 0 to 100, a higher score refers to higher body resources.

CONTACTS AND LOCATIONS:
Overall Officials: Katriina Hyvönen, PhD, Principal Investigator — JAMK University Of Applied Sciences
Locations (1):
- JAMK University of Applied Sciences, Jyväskylä, Finland

IPD SHARING:
Plan to Share IPD: Yes
Data from surveys and physiological measurements will be anonymised after the research and will be archived to the research data storage service (IDA). Anonymised data will open for reuse after the research finishes in 2024. The reuse of interview data will be restricted to suitable parts.
Supporting Information: Study Protocol